CLINICAL TRIAL: NCT03715868
Title: Pre-operative Short-term Administration of a Formula Diet Containing a Non-milk-derived Protein Source for Prevention of Acute Kidney Injury After Cardiac Surgery
Acronym: UNICORN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Volker Burst, Medical Doctor, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 004
Record Dates: First submitted 2018-10-11; First posted 2018-10-23 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Acute Renal Failure; Acute Kidney Injury
Keywords: Acute kidney injury; Acute renal failure; Diet; Cardiothoracic surgery; Change of protein source
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-milked derived protein source formula diet (Active Comparator): Formula diet based on a non-milked derived protein source
  Interventions: Other: Non-milked derived protein source formula diet
- Milked derived protein source formula diet (No Intervention): Formula diet based on a milked derived protein source

INTERVENTIONS:
Other: Non-milked derived protein source formula diet — Formula diet based on a non-milked derived protein source
  Arms: Non-milked derived protein source formula diet

SUMMARY:
Cardiac surgery is associated with a high risk of postoperative AKI with significant morbidity and mortality. To date, no preventive or therapeutic measures exist to prevent this. According to the data from animal trials, a preoperative diet with a deficiency of milk-derived proteins may be a new preventive measure in this context.

This trial will investigate whether one week of changing the diets protein source to a non-milk-derived one prior to surgery effectively induces renal protection from post-surgery AKI in humans. Patients undergoing elective cardiac surgery are randomized into two arms. In the non-milked-derived based diet arm, patients receive an appropriate formula diet based on a protein source other than milk derived proteins. In the control arm, patients are provided with a formula diet based on milk-protein. Total amount of calories and proteins is not restricted and - due to randomization - assumed not to be significantly different between the two arms.

DETAILED DESCRIPTION:
Cardiac surgery is associated with a high risk of postoperative AKI with significant morbidity and mortality. Acute kidney injury (AKI) constitutes a significant complication in hospitalized patients with an incidence of about 30%. Depending on existing comorbidities, a mortality of up to 60% occurs in critically ill or postoperative patients with AKI. To date, no preventive or therapeutic measures exist to prevent this. According to the data from animal trials, a preoperative diet low in sulfur-containing amino acids may be a new preventive measure in this context.

This trial will investigate whether one week of changing the diets protein source to a non-milk-derived one prior to surgery effectively induces renal protection from post-surgery AKI in humans. Patients undergoing elective cardiac surgery are randomized into two arms.

In the non-milked-derived based diet arm, patients receive an appropriate formula diet based on a protein source other than milk derived proteins. The formula diet replaces the regular diet completely from day -7 until the scheduled cardiothoracic surgery. The amount of formula diet is based on individual calculations to cover the patients daily energy demand.

In the control arm, patients are provided with a formula diet based on milk-protein, accordingly. Total amount of calories and proteins is not restricted and - due to randomization - assumed not to be significantly different between the two arms.

The primary endpoint of the clinical trial is to investigate whether a preoperative diet with a deficiency of milk-derived proteins leads to a reduction of AKI incidence within 72 hours after surgery. AKI is defined according to 'Kidney Disease: Improving Global Outcomes' (KDIGO) classification as an increase in serum creatinine of ≥0.3 mg/dl within 48 hours, or an increase of serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days, or a reduction of urine output to <0.5ml/kg/hour for more than 6 hours.

Baseline creatinine will be assessed prior to the start of the surgical procedure. The time frame for the following assessments with respect to the primary endpoint will be 72 hours from the onset of ischemia (cross-clamping). Blood samples will be obtained at 24 hours, 48 hours, and 72 hours after cross-clamping. Hourly urine output will be assessed as long as a Foley-catheter is in place.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥50 years of age
2. Caucasian ethnicity
3. Scheduled cardiac surgery with use of the heart-lung machine with a lead time of at least 9 days
4. Written informed consent

Exclusion Criteria:

1. Chronic renal replacement therapy
2. Status post kidney transplantation
3. Vegetarian lifestyle
4. BMI <18.5 kg/m2
5. Calorie-reduced diet within the preceding 4 weeks
6. Underlying wasting disease
7. Uncontrolled local or systemic infection
8. Contraindication for enteral nutrition
9. Known allergy to or intolerance of the ingredients of the formula diets used
10. Pregnancy or breastfeeding
11. Absence of safe contraceptive measures or non-occurrence of menopause (in women)
12. Participation in other interventional trials
13. Persons who are in a dependency/employment relationship with the investigators
14. Accommodation in an institution by judicial or administrative order.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
AKI incidence within 72 hours according KDIGO classification after induction of ischemia ('cross clamping') in comparison to baseline values | Pre-operative baseline day of surgery to 72 hours after induction of ischemia
  The primary endpoint of the clinical trial is to investigate whether a preoperative diet with a non-milked derived protein source leads to a reduction of AKI incidence within 72 hours after surgery. AKI is defined according to KDIGO as an increase in serum creatinine of ≥0.3 mg/dl within 48 hours, or an increase of serum creatinine to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days, or a reduction of urine output to <0.5ml/kg/hour for more than 6 hours.
  Baseline creatinine will be assessed prior to the start of the surgical procedure. The time frame for the following assessments with respect to the primary endpoint will be 72 hours from the onset of ischemia (cross-clamping). Blood samples will be obtained at 24 hours, 48 hours, and 72 hours after cross-clamping. Hourly urine output will be assessed as long as a Foley-catheter is in place.

SECONDARY OUTCOMES:
Absolute and relative increase of serum creatinine concentration at 24 hours, 48 hours, and 72 hours after cardiac surgery ("cross clamping") | Pre-operative baseline day of surgery and 24 hours, 48 hours and 72 hours after induction of ischemia
Incidence of AKI as defined by KDIGO until discharge | Pre-operative baseline day of surgery to day of discharge, an expected average of 10 days
Occurrence of AKI according to KDIGO I, II, III | Pre-operative baseline day of surgery to day of discharge, an expected average of 10 days
Maximum serum creatinine concentration detected postoperatively during hospitalization | Pre-operative baseline day of surgery to day of discharge, an expected average of 10 days
Need for renal replacement treatment during hospitalization | Patient will be followed up for the duration of hospital stay, an expected average of 10 days
In-hospital mortality | Patient will be followed up for the duration of hospital stay, an expected average of 10 days
Length of hospital stay | Patient will be followed up for the duration of hospital stay, an expected average of 10 days
Length of stay on intensive care unit (ICU) | Day of admittance until day of discharge from ICU, an expected average of 2 days
tissue inhibitor of metalloproteinases 2 (TIMP-2) and insulin-like growth factor-binding protein 7 (IGFBP7) urine concentrations before surgery and at 4 hours and 24 hours after onset of ischemia (NephroCheck Test) | Pre-operative baseline day of surgery and at 4 hours and 24 hours after induction of ischemia
C-reactive Protein (CRP) concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
Leukocyte count | Pre-operative day of surgery and at 24 hours after onset of ischemia
Creatine kinase concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
Troponin T concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
Lactate Dehydrogenase concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
N-terminal Pro brain natriuretic peptide (NT-ProBNP) concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
Lactate concentration | Pre-operative day of surgery and at 24 hours after onset of ischemia
Amino acid pattern (concentrations), Insulin concentration, insulin-like growth factors (IGF1) concentration, glucose concentration | Before start of diet and on day of admission (before surgery)
Mortality rate at 30 and 180 days (as followed-up upon by telephone call) | Day of surgery until 180 days after time point of surgery
Need for renal replacement therapy within 180 days after time point of surgery (as followed-up upon by telephone call) | Day of surgery until 180 days after time point of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Osterholt T, Gloistein C, Todorova P, Becker I, Arenskrieger K, Melka R, Koehler FC, Faust M, Wahlers T, Benzing T, Muller RU, Grundmann F, Burst V. Preoperative Short-Term Restriction of Sulfur-Containing Amino Acid Intake for Prevention of Acute Kidney Injury After Cardiac Surgery: A Randomized, Controlled, Double-Blind, Translational Trial. J Am Heart Assoc. 2022 Sep 6;11(17):e025229. doi: 10.1161/JAHA.121.025229. Epub 2022 Sep 3. PMID 36056721